CLINICAL TRIAL: NCT01842945
Title: Internet Based Cognitive Behavior Therapy for Procrastination: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCT01842945; 2011-38394-87877-7 (Other Grant/Funding Number: Swedish Research Council)
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Procrastination
Keywords: Procrastination; internet based cognitive behavior therapy; randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wait-list control (No Intervention)
- Treatment with therapist contact (Experimental)
  Interventions: Behavioral: Internet-based cognitive behavioural therapy (iCBT) with therapist contact.
- Treatment without therapist contact (Experimental)
  Interventions: Behavioral: Internet-based cognitive behavioural therapy (iCBT) without therapist contact.

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioural therapy (iCBT) without therapist contact. — The iCBT consists of our structured self-help program lasting a total of eight active treatment weeks and does not include a therapist contact.
  Arms: Treatment without therapist contact
Behavioral: Internet-based cognitive behavioural therapy (iCBT) with therapist contact. — The iCBT consists of our structured self-help program lasting a total of eight active treatment weeks and includes a therapist contact.
  Arms: Treatment with therapist contact

SUMMARY:
The aim of this study is to examine the effects of cognitive behavior therapy (CBT) for procrastination, and to investigate whether it can be delivered via the Internet. Two treatment groups will be used, one with therapist contact and one without, as well as a wait-list control group. It is assumed that the treatment group with therapist contact will be superior to the treatment group receiving no therapist contact since procrastination can be partially explained as a self-regulatory failure. Both treatment groups are presumed to be superior to the wait-list control.

ELIGIBILITY:
Inclusion Criteria:

* Primary difficulties are caused by chronic and severe procrastination
* Swedish residency
* Fluent in Swedish
* Computer with internet access

Exclusion Criteria:

* Ongoing psychotherapy
* Ongoing psychotropic medication (unless stabilized for three months)
* Severe depression (> 30 points on MADRS-S)
* Suicidal ideation
* Misuse of drugs or alcohol
* Bipolar disorder
* Schizophrenia or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pure Procrastination Scale (PPS) | 0 weeks and 10 weeks
  The PPS features twelve items measuring the prevalence of procrastination.
Change from baseline in Pure Procrastination Scale (PPS) | 0 weeks and 60 weeks
  The PPS features twelve items measuring the prevalence of procrastination.
Change from baseline in Susceptibility to Temptation Scale (STS) | 0 weeks and 10 weeks
  The STS features eleven items measuring the susceptibility to temptation, which can affect the ability to follow through a task or commitment.
Change from baseline in Susceptibility to Temptation Scale (STS) | 0 weeks and 60 weeks
  The STS features eleven items measuring the susceptibility to temptation, which can affect the ability to follow through a task or commitment.
Change from baseline in Irrational Procrastination Scale (IPS) | 0 weeks and weekly during treatment period of 10 weeks
  The IPS features nine items measuring the degree of irrational delay causing procrastination.
Change from baseline in Irrational Procrastination Scale (IPS) | 0 weeks and 60 weeks
  The IPS features nine items measuring the degree of irrational delay causing procrastination.

SECONDARY OUTCOMES:
Change from baseline in Montgomery Asberg Depression Rating Scale Self-report version (MADRS-S) | 0 weeks and 10 weeks
  MADRS-S is a self-assessment version of MADRS and features nine items measuring changes in mood, anxiety, sleeping patterns, appetite, concentration, initiative, emotional engagement, pessimism and attitude towards life.
Change from baseline in Montgomery Asberg Depression Rating Scale Self-report version (MADRS-S) | 0 weeks and 60 weeks
  MADRS-S is a self-assessment version of MADRS and features nine items measuring changes in mood, anxiety, sleeping patterns, appetite, concentration, initiative, emotional engagement, pessimism and attitude towards life.
Change from baseline in Generalized Anxiety Disorder Assessment 7-item (GAD-7) | 0 weeks and 10 weeks
  GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Change from baseline in Generalized Anxiety Disorder Assessment 7-item (GAD-7) | 0 weeks and 60 weeks
  GAD-7 features seven items for assessing anxiety and screening for generalized anxiety disorder.
Change from baseline in Quality of Life Inventory (QOLI) | 0 weeks and 10 weeks
  QOLI features 32 items concerning 16 areas of life rated by the subject concerning importance and satisfaction.
Change from baseline in Quality of Life Inventory (QOLI) | 0 weeks and 60 weeks
  QOLI features 32 items concerning 16 areas of life rated by the subject concerning importance and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Study Director — Stockholm University
Locations (1):
- Department of Psychology, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rozental A, Carlbring P. Internet-based cognitive behavior therapy for procrastination: study protocol for a randomized controlled trial. JMIR Res Protoc. 2013 Nov 12;2(2):e46. doi: 10.2196/resprot.2801. PMID 24220277
- [Background] Rozental A, Forsell E, Svensson A, Andersson G, Carlbring P. Overcoming procrastination: one-year follow-up and predictors of change in a randomized controlled trial of Internet-based cognitive behavior therapy. Cogn Behav Ther. 2017 Apr;46(3):177-195. doi: 10.1080/16506073.2016.1236287. Epub 2016 Sep 29. PMID 27682415
- [Result] Rozental A, Forsell E, Svensson A, Andersson G, Carlbring P. Internet-based cognitive-behavior therapy for procrastination: A randomized controlled trial. J Consult Clin Psychol. 2015 Aug;83(4):808-24. doi: 10.1037/ccp0000023. Epub 2015 May 4. PMID 25939016
- [Derived] Rozental A, Forsell E, Svensson A, Forsstrom D, Andersson G, Carlbring P. Psychometric evaluation of the Swedish version of the pure procrastination scale, the irrational procrastination scale, and the susceptibility to temptation scale in a clinical population. BMC Psychol. 2014 Dec 11;2(1):54. doi: 10.1186/s40359-014-0054-z. eCollection 2014. PMID 25566392